CLINICAL TRIAL: NCT06649188
Title: Electromotive Drug Administration of Magnesium Sulphate on Hypertrophic Scar Post-Burn
Brief Title: Electromotive Drug Administration of Magnesium Sulphate on Hypertrophic Scar
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Gamal Fawzy El-Sayed, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005334
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Hypertrophic Scars
Keywords: Iontophoresis; Post burn
MeSH Terms: conditions — Cicatrix, Hypertrophic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Magnesium Sulphate Iontophoresis (Experimental)
  Interventions: Device: Magnesium Sulphate Iontophoresis; Other: traditional physical therapy program
- Group B: Control (Sham Comparator)
  Interventions: Other: traditional physical therapy program

INTERVENTIONS:
Device: Magnesium Sulphate Iontophoresis — Iontophoretic drug delivery system (phoresors II auto model PM850 IOMED) The phoresors II auto model PM850 IOMED allows the user to deliver a specific dose from 0 to 80 mA/min, control the current from 0 to 4 mA and automatically calculates required time for the selected dose. Current ramp-up and down, shut-off, error messages and safety checks are also performed automatically. The builtin option for manual current shut-off is an added safety feature (Teslim et al., 2013).
  * Electrodes: Active-Anode (Drug Delivery).
  * Drug Used: MgSO4 Aqueous Solution.
  * Drug Ion Polarity: Positive Polarity.
  Arms: Group A: Magnesium Sulphate Iontophoresis
Other: traditional physical therapy program — Deep friction massage, stretching and pressure therapy.

SUMMARY:
In this study 80 patients will be randomly assigned into two equal groups (40 patients for each group):

1. Group A: Experimental: Magnesium Sulphate Iontophoresis for Postburn Hypertrophic Scar The study group includes 40 postburn hypertrophic scar patients will receive Magnesium Sulphate iontophoresis twice a week for 4 weeks; in addition to their traditional physical therapy program (deep friction massage, stretching and pressure therapy).
2. Group B: Control: Traditional physical therapy for postburn hypertrophic scar This group includes 40 patients with postburn hypertrophic scar who will receive only the traditional PT (deep friction massage, stretching and pressure therapy) 2 sessions per week for 4 weeks

DETAILED DESCRIPTION:
1. Assessment measures and procedures:

   1. High resolution ultrasonography [Time Frame: Change of hypertrophic scar thickness from the beginning of treatment to the end of treatment (after 4 and 12 weeks from the beginning of treatment).

      High frequency ultrasound is the most common used technique for scar assessment. Its inferior resolution compared to optical equivalents is mitigated by its superior penetration depth allowing thickness analysis, even in severe scar thickening. The working mechanism is based on refection of sound waves of structures with different acoustic impedances and the analysis of the refection time to determine the depth of the structure. The penetration depth ranges from the upper dermal layers to full-thickness skin and subcutaneous structures, depending on the employed frequency (Elrefaie et al., 2020).
   2. Patient and observer scar assessment scale [Time Frame: Assessing the change of patient and observer scar assessment scale score from baseline (beginning of treatment) to 4 and 12 weeks after treatment.

   The scar will be rated numerically on a ten-step scale by both the patient and doctor on six items: vascularity, pigmentation, thickness, relief, pliability, and surface area on the Observer Scale. The Patient Scale consists of pain, itchiness, color, stiffness, thickness, and irregularity of the scar. Minimal score means good progression and maximum score means the scare is worse (Lenzi et al., 2019).
2. Treatment procedures:

Iontophoretic drug delivery system (phoresors II auto model PM850 IOMED) The phoresors II auto model PM850 IOMED allows the user to deliver a specific dose from 0 to 80 mA/min, control the current from 0 to 4 mA and automatically calculates required time for the selected dose. Current ramp-up and down, shut-off, error messages and safety checks are also performed automatically. The builtin option for manual current shut-off is an added safety feature (Teslim et al., 2013).

* Electrodes: Active-Anode (Drug Delivery).
* Drug Used: MgSO4 Aqueous Solution.
* Drug Ion Polarity: Positive Polarity. Prior to intervention, skin sensation will be assessed using warm water in a test-tube (temperature), pin prick (pain) and cotton wool (light touch) to ascertain the skin sensitivity.

Before each treatment, the surface area of the scar will be cleaned with cotton wool and alcohol to reduce skin resistance. 2.5 ML MgSO4 will be applied to the active positive electrode via a syringe with concentration 100 mg/cm2 (it's available in hospitals and not found in pharmacies), active electrode will be placed directly over the hypertrophic scar. The dispersive electrode will be applied to the skin 6 inch distal from the active electrode (Evans et al., 2001).

The dose needed will be selected in the device which is 75 mA/min (Teslim et al., 2013) then the current will be increased gradually depending on subject tolerance, ranging from 2 to 4 mA, the device will automatically calculate the required time for the selected dose. The interventions will be repeated twice a week for 4 weeks (Teslim et al., 2013). If a subject reports any sensation other than tingling, the treatment will be stopped, the electrodes will be removed and the skin will be inspected (Evans et al., 2001).

ELIGIBILITY:
Inclusion Criteria:

* 1-Patient with hypertrophic scar (3-6) months after burn healing. 2-Age range between 20-40 years. 3-Male and female patients will participate in the study. 4-All patients have a post-burn hypertrophic scar at different body sites. 5-All patients enrolled on the study will have their informed consent.

Exclusion Criteria:

- 1-Patients with prior medical histories of cardiac arrhythmias. 2-Patients with cardiac pacemakers. 3-Patients with orthopaedic implants. 4-Areas of skin with lesions and impaired sensation. 5-During pregnancy and breastfeeding. 6-Patient with diabetes mellitus. 7-Patients with a history of hypersensitivity or adverse reactions associated with (MgSO4).

8-Recent MgSO4 administration 6 months before the study. 9-Any subject complaining of psychiatric disorders or neurological disorders such as myasthenia gravis

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Change of hypertrophic scar thickness | 4 weeks
  High frequency ultrasound is the most common used technique for scar assessment. Its inferior resolution compared to optical equivalents is mitigated by its superior penetration depth allowing thickness analysis, even in severe scar thickening. The working mechanism is based on refection of sound waves of structures with different acoustic impedances and the analysis of the refection time to determine the depth of the structure. The penetration depth ranges from the upper dermal layers to full-thickness skin and subcutaneous structures, depending on the employed frequency (Elrefaie et al., 2020).
The change of patient and observer scar assessment scale score | 4 weeks
  The scar will be rated numerically on a ten-step scale by both the patient and doctor on six items: vascularity, pigmentation, thickness, relief, pliability, and surface area on the Observer Scale. The Patient Scale consists of pain, itchiness, color, stiffness, thickness, and irregularity of the scar. Minimal score means good progression and maximum score means the scare is worse (Lenzi et al., 2019).

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt